## INFROMED CONSENT FOR PARTICIPATION IN AN OBSERVATIONAL STUDY

«Rehabilitation of the patients recovered from the pneumonia associated with the novel COVID-19 infectious disease»

Approval Number 145 by Ethical Board as of 09/16/2020.

## INFROMED CONSENT FOR PARTICIPATION IN AN OBSERVATIONAL STUDY

«Rehabilitation of the patients recovered from the pneumonia associated with the novel COVID-19 infectious disease»

I am familiar with the results of my previous medical examinations including laboratory investigation of the presence of SARS-CoV-2 RNA, multi-spiral CT of the lungs, and the medical conclusions of the doctors conducted treatment of my COVID-19 pulmonary infection. I am informed that after the SARS-CoV-2 pneumonia I may experience such symptoms as increased fatigue, malaise, shortness of breath, racing of the heart during routine physical activity. Moreover, it was clarified to me that the novel COVID-19 infectious disease may cause damage of the cardiovascular system (Outcomes of Cardiovascular Magnetic Resonance Imaging in Patients Recently Recovered from Coronavirus Disease 2019. JAMA, Cardiol. doi:10.1001/jamacardio.2020.3557; Temporary recommendations "Prophylaxis, diagnostics, and treatment of novel COVID-19 infectious disease", version 7 (6/3/2020) Healthcare Ministry of the Russian Federation).

I consent to take a part in an observational study of the patients recovered from the COVID-19 associated pneumonia. This study will take place at Autonomous Healthcare Institution of Voronezh Region "Voronezh Region Clinical, Consultative and Diagnostic Center" and will be conducted by the certified medical specialists, primarily lung specialists and cardiologists.

I consent to provide my medical history, complete questionnaires, and undergo the workup of my blood samples (total volume of 15-20 cc) to evaluate the inflammatory level, lipid and glycemic profiles, kidney and liver functions, and also level of the specific cardiac markers.

According to the specialists' recommendations I may undertake electrocardiography, heart ultrasound, heart magnetic tomography with contrast which will be injected intravenously (this will be explained additionally before the procedure), multi-spiral computed tomography of the lungs, evaluation of the lung functions, and other investigations in case of need in accordance to my current health state. Based on the results of the examinations I will be advised on the specific physical regimen, dietary recommendations, lifestyle modifications, pharmacological therapy aimed to respiratory and cardiovascular recovery in a strict compliance with the clinical recommendations and current guidelines. As a part of this study, observation is conducted at Autonomous Healthcare Institution of Voronezh Region "Voronezh Region Clinical, Consultative and Diagnostic Center" with the planned 2-3 follow up visits in the period of 12 months.

I consent that the medical doctors engaged in this study may inform my family members regarding my diseases and general health state.

I understand that all the documentation with my personal identification will be handled in a strict confidentiality in accordance to the current jurisdiction and government laws. I also understand that in case of publication of this study in medical nomenclature my personal data and identification information will not be disclosed.

I have fully read this informed consent, am completely aware of the specifics of this study, and agree with its importance. I have discussed all the questions regarding my health with the doctor and I agree to voluntarily participate in this observational study while following all the needed medical recommendations.

| Patient's name | | | (Name and Surname) |
|---------------------|----------|-----------------|--------------------|
| Patient's signature | <u> </u> | | 20 |
| Doctor's name | | | (Name and Surname) |
| Doctor's signature | <b>«</b> | <b>&gt;&gt;</b> | 20 |